CLINICAL TRIAL: NCT05583877
Title: DM-BOOST Para Latinx: a Diabetes Mellitus Program Using Behavioral Economics to Optimize Outreach and Self-management Support With Technology for Latinx Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Amante (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Daniel Amante, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00000376; 1K01DK131318 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to culturally-adapt a patient-centric intervention designed to improve implementation of diabetes self-management training in Spanish-speaking patients. To accomplish cultural adaptation of the DM-BOOST intervention, a Patient Research Expert Panel (PREP) (n</=4) will participate in Community Engagement Studios to inform adaptations (Aim 1) and usability test the intervention (Aim 2). A randomized pilot with new patients (n</=70) will then be conducted to assess feasibility (Aim 3).
Who Masked: Participant, Investigator
Masking Description: After completing the informed consent, study staff will enter the participant's information into pre-populated REDCap identification numbers. This will assign allocation based on the randomization table. Using this technique, participants will be blinded to allocation. However, research staff will not be blinded to provide personalized training for intervention and control. The investigator will be blinded to randomization for all participants during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Diabetes BOOST (Experimental): Intervention group participants will complete a baseline survey, receive a referral to DSMT from the research team, a mailed welcome letter and self-care education sent via a series of personalized patient portal secure messages, text messages, and video call. They will be sent text messages with information about one of the American Association of Diabetes Educators 7 self-care behaviors and will receive encouragement to author their own self-management behavioral goals. Participants will also complete a telehealth training video call with research staff to review the functionality of their patient portal and refine diabetes-related goals. The participant will then be encouraged to send a patient portal message to their DSMT CDCES that includes their personalized goals prior to their scheduled DSMT session. They will then complete a 3-month follow-up survey and qualitative interview.
  Interventions: Behavioral: Diabetes BOOST
- Usual Care (Active Comparator): Comparison Group participants will complete a baseline survey, receive a DSMT referral request from research team to their primary care provider and a mailed welcome letter. The mailed letter will welcome the participant to the study and contain general information about diabetes self-care behaviors and goal setting. They will complete a DSMT session. They will then complete a 3-month follow-up survey and qualitative interview.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Diabetes BOOST — Participants will receive supportive care using technology for DSMT in addition to usual care.
  Arms: Intervention - Diabetes BOOST
Behavioral: Usual Care — Participants will receive usual care for DSMT.
  Arms: Usual Care

SUMMARY:
The specific aims of this project are to culturally adapt the DM-BOOST intervention for Latinx patients, usability test 'DM-BOOST para Latinx' to optimize cultural appropriateness and patient engagement and conduct a feasibility evaluation of DM-BOOST para Latinx. These aims will be accomplished via a community-based participatory research approach in collaboration with clinical, community and patient partners. This project will inform subsequent proposals to evaluate implementation of DM-BOOST in the UMass Memorial Health Care system.

ELIGIBILITY:
Aims 1 and 2 Patient Inclusion Criteria:

* Age > 18 years
* Diagnosis of type 2 diabetes
* Identifies as Hispanic/Latinx
* Spanish language preference

Aims 1 and 2 Patient Exclusion Criteria:

* Cognitive impairment
* Current prisoner
* Pregnant women

Aim 3 Patient Inclusion Criteria:

* Age > 18 years
* Diagnosis of type 2 diabetes
* Identifies as Hispanic/Latinx
* Spanish language preference

Aim 3 Patient Exclusion Criteria:

* Cognitive impairment
* Current prisoner
* Pregnant women
* Completed DSMT in previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Process Evaluation | 3 - 6 months
  Evaluate engagement by examining the number of DSMT appointments scheduled, cancellation/no show rates and total number of DSMT-related encounters completed.

SECONDARY OUTCOMES:
Diabetes self-efficacy | 3 months
  Diabetes self efficacy will be measured at baseline and 3 months after enrolling in the study using the Diabetes Management Self-Efficacy Scale. Participants will provide feedback on set of questions, using a 5-point Likert scale( with 1=Strong Disagree, 2=Somewhat Disagree, 3= Neutral, 4=Somewhat Agree, 5= Strongly Agree)
Diabetes treatment satisfaction | 3 months
  Diabetes Treatment Satisfaction will be measured at 3 months after enrolling in the study using the Diabetes Treatment Satisfaction Questionnaire Change tool. Participants will be asked to share how their experience of current treatment has changed from their experience of treatment before the study began. They will answer each question by choosing 3 for Much More Satisfied Now up to -3 for Much Less Satisfied Now. (3,2,1,0,-1,-2,-3)
Change in HbA1c Percentage | 6 months
  Measurement of HbA1c values to determine impact of intervention. HbA1c values at baseline visit will be compared with values at 3-6 months after participant's enrollment. These data will be obtained through EHR chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Amante, PhD, MPH, Principal Investigator — UMass Chan Medical School
Locations (2):
- United States (2):
  - UMass Memorial health, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No